CLINICAL TRIAL: NCT06822790
Title: A Phase 3 Open-Label Extension Study to Evaluate the Long-Term Safety and Efficacy of Plozasiran in Adults With Hypertriglyceridemia (SHASTA-10 Study)
Brief Title: Long-Term Safety and Efficacy of Plozasiran in Adults With Hypertriglyceridemia
Acronym: SHASTA-10
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AROAPOC3-3006
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — plozasiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Plozasiran Injection (Experimental): 8 doses of plozasiran (ARO-APOC3) administered by subcutaneous (SC) injection
  Interventions: Drug: Plozasiran Injection

INTERVENTIONS:
Drug: Plozasiran Injection — ARO-APOC3 injection
  Other Names: ARO-APOC3

SUMMARY:
This is an open-label study to be conducted in adults with hypertriglyceridemia (HTG) and severe hypertriglyceridemia (SHTG). Each participant must have completed all required visits per protocol in the parent study AROAPOC3-2003 (USA and Canada participants only; NCT# 05413135), AROAPOC3-3001(Canada and Japan participants only; NCT05089084), AROAPOC3-3003 (NCT06347003), AROAPOC3-3004 (NCT06347016) or AROAPOC3-3009 (Argentina, Italy, South Africa, and Spain; NCT06347133).

Subjects who previously met all eligibility requirements for AROAPOC3-3003 or AROAPOC3-3004 and were not permitted to proceed to randomization per the Sponsor's direction in order to prevent excessive over-enrollment may also be enrolled in this trial. The subjects must meet all other applicable eligibility criteria prior to enrollment and have an HbA1c results of <=10% within 30 days prior to Day 1.

Subjects entering this OLE from AROAPOC3-2003 must meet the following additional criteria to be considered for enrollment in addition to applicable eligibility criteria:

1. HbA1c ≤10% within 30 days prior to Day 1
2. Completed AROAPOC3-2001 prior to entry into AROAPOC3-2003 AND fulfill either (c) or (d)
3. Baseline fasting TG level of ≥500 mg/dL and prior history of acute pancreatitis at the time of enrollment into AROAPOC3-2001
4. Baseline fasting TG level of ≥1000 mg/dL at the time of enrollment into AROAPOC3-2001

All eligible participants will receive plozasiran administered subcutaneously (SC) approximately every 3 months for 24 months. Participants will be counseled to remain on the specified low-fat diet throughout the study in accordance with local standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Adult males, or nonpregnant (who do not plan to become pregnant), nonlactating adult females, who are able and willing to provide written informed consent prior to the performance of any study-specific procedures
* Completed all required study visits per protocol in the parent study
* Female subjects of childbearing potential must agree to use a highly effective method of contraception during the study and for at least 90 days after the End of Study (EOS) or the last dose of plozasiran, whichever is later. Male subjects must agree to use a condom during the study and for at least 90 days after the EOS or last dose of plozasiran whichever is later. Subjects must not donate sperm or eggs during the study and for at least 90 days after the EOS or last dose of plozasiran, whichever is later. Female subjects of childbearing potential on hormonal contraceptives must be stable on medication for >1 menstrual cycle prior to Day 1.
* Subjects must be on standard of care lipid and TG-lowering medications per local guidelines (unless documented as intolerant as determined by the Investigator, including an inability to safely administer or re-administer a specific drug because of fear, preference, genetic, clinical, or metabolic considerations, or due to a previous adverse reaction associated with, attributed to, or caused by specific drug)
* If the subject has a medical history of clinical atherosclerotic cardiovascular disease (ASCVD) or elevated 10-year ASCVD risk (eg, ≥7.5% per American Heart Association/American College of Cardiology [AHA/ACC] risk calculator for subjects ≥40 years of age or Framingham risk score calculator for subjects under the age of 40), the subject must be on appropriate lipid-lowering therapy as per local standard of care (ie, including moderate-to-high intensity statin, as indicated).

If the subject has diabetes:

1. Subject must be on optimized antidiabetic regimen as defined by the local standards, Investigator, and institutional practices
2. Subject must have no events of diabetic ketoacidosis, diabetic decompensation/ hyperosmolar hyperglycemic nonketotic coma, diabetes complications, recurrent infections, or hospitalization related to poor glycemic control within 24 weeks of the Day 1 visit - Willing to follow diet counseling and maintain a stable low-fat diet

Subjects in the USA and Canada who completed protocol AROAPOC3-2003 meeting all eligibility criteria (with the exception of inclusion criteria #9 which is not applicable to these subjects) who also meet the following additional criteria may enroll in this trial:

* HbA1c ≤10% within 30 days prior to Day 1
* Completed AROAPOC3-2001 prior to entry into AROAPOC3-2003 AND either (c) or (d) below:
* Baseline fasting TG level of ≥500 mg/dL and prior history of acute pancreatitis at the time of enrollment into AROAPOC3-2001
* Baseline fasting TG level of ≥1000 mg/dL at the time of enrollment into AROAPOC3-2001

  * Subjects who previously met all eligibility requirements for AROAPOC3-3003, or AROAPOC3-3004 and were not permitted to proceed to randomization per Sponsor's direction in order to prevent excessive over-enrollment may also be enrolled in this trial. These subjects must meet all eligibility criteria prior to enrollment (with the exception of inclusion criteria #2 and #8 which are not applicable to these subjects) and have an HbA1c ≤10% within 30 days of Day 1.

Exclusion Criteria:

* Subject was permanently discontinued from receiving plozasiran in the parent study due to elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) or due to HbA1c elevation that did not respond to antidiabetic regimen
* Subject withdrew consent for continued study treatment in the parent study
* Known hypersensitivity to the active substance or to any of the excipients of plozasiran
* Known hypersensitivity to the active substance or to any of the excipients of plozasiran
* Any new condition or worsening of existing condition or any other situation that in the Investigator's judgment, would make the subject unsuitable for enrollment, could interfere with the subject participating in or completing the study, would make it difficult to comply with protocol requirements, or put the subject at an additional safety risk
* Unwilling to limit alcohol consumption to within moderate limits for the duration of the study.
* Poorly controlled glycemia (ie, HbA1c >10%) based upon the most recent HbA1c level reported in the parent trial prior to Day 1
* Acute pancreatitis within 4 weeks prior to Day 1
* Use of any hepatocyte-targeted siRNA that targets lipids and/or triglycerides within 365 days before Day 1 (except plozasiran or inclisiran, which are permitted). Administration of inclisiran must be separated from administration of plozasiran by at least 4 weeks throughout the treatment period
* Use of any other hepatocyte targeted siRNA or antisense oligonucleotide molecule within 60 days or within 5 half-lives before Day 1 based on plasma PK, whichever is longer.
* Use of an investigational agent (other than plozasiran) or device within 30 days or within 5 half-lives, based on plasma PK, whichever is longer, prior to Day 1 (V1) or current participation in an interventional investigational study.
* Recent unstable or symptomatic cardiac arrhythmia (including any associated medication changes) within 90 days prior to Day 1. Individuals with stable well-controlled atrial arrhythmias will be allowed to participate in the study.
* Uncontrolled hypertension (ie, seated systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg) at Day 1; subject may be re-evaluated when hypertension is controlled.

Note: Other inclusion/exclusion criteria may apply per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 869 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | From first dose of study drug through Month 24

SECONDARY OUTCOMES:
Change from Baseline Over Time in Fasting Serum Triglyceride (TG) Levels | From first dose of study drug through Month 24
Percent Change from Baseline Over Time in Fasting Serum TG Levels | From first dose of study drug through Month 24
Change from Baseline Over Time in Apolipoprotein CIII (APOC3) | From first dose of study drug through Month 24
Percent Change from Baseline Over Time in APOC3 | From first dose of study drug through Month 24
Change from Baseline Over Time in Remnant Cholesterol | From first dose of study drug through Month 24
Percent Change from Baseline Over Time in Remnant Cholesterol | From first dose of study drug through Month 24
Change from Baseline Over Time in Fasting Non-High-Density Lipoprotein Cholesterol (non-HDL-C) | From first dose of study drug through Month 24
Percent Change from Baseline Over Time in Fasting non-HDL-C | From first dose of study drug through Month 24
Change from Baseline Over Time in Fasting High-Density Lipoprotein Cholesterol (HDL-C) | From first dose of study drug through Month 24
Percent Change from Baseline Over Time in Fasting HDL-C | From first dose of study drug through Month 24
Change from Baseline Over Time in Fasting Total Apolipoprotein B (Apo B) | From first dose of study drug through Month 24
Percent Change from Baseline Over Time in Fasting Total Apo B | From first dose of study drug through Month 24
Change from Baseline Over Time in Fasting Low-Density Lipoprotein Cholesterol (LDL-C) using Ultracentrifugation | From first dose of study drug through Month 24
Percent Change from Baseline Over Time in Fasting LDL-C using Ultracentrifugation | From first dose of study drug through Month 24
Change from Baseline Over Time in Hemoglobin A1c (HbA1c) | From first dose of study drug through Month 24
Number of Participants With Emergent Apheresis | From first dose of study drug through Month 24
Adjudicated Major Adverse Cardiovascular Event Rates During the Treatment Period | From first dose of study drug through Month 24
Incidence of Anti-Drug Antibodies (ADA) to Plozasiran Over Time | From first dose of study drug through Month 24
Titers of ADA to Plozasiran Over Time | From first dose of study drug through Month 24
Adjudicated Acute Pancreatitis (AP) Event Rate During the Treatment Period | From first dose of study drug through Month 24

CONTACTS AND LOCATIONS:
Locations (39):
- United States (33):
  - Research Site 21, Bakersfield, California
  - Research Site 9, Beverly Hills, California
  - Research Site 11, Canoga Park, California
  - Research Site 39, Lincoln, California
  - Research Site 34, Oxnard, California
  - Research Site 14, Hialeah, Florida
  - Research Site 1, Miami Lakes, Florida
  - Research Site 38, North Miami, Florida
  - Research Site 16, Tamarac, Florida
  - Research Site 18, Tampa, Florida
  - Research Site 17, Park Ridge, Illinois
  - Research Site 28, Overland Park, Kansas
  - Research Site 23, Topeka, Kansas
  - Research Site 12, Annapolis, Maryland
  - Research Site 30, Flint, Michigan
  - Research Site 33, Jackson, Mississippi
  - Research Site 32, Olive Branch, Mississippi
  - Research Site 2, Jefferson City, Missouri
  - Research Site 29, Fremont, Nebraska
  - Research Site 3, Omaha, Nebraska
  - Research Site 37, Asheboro, North Carolina
  - Research Site 36, Morehead City, North Carolina
  - Research Site 22, Beavercreek, Ohio
  - Research Site 31, Oklahoma City, Oklahoma
  - Research Site 26, Horsham, Pennsylvania
  - Research Site 8, Newport, Pennsylvania
  - Research Site 27, El Paso, Texas
  - Research Site 24, Houston, Texas
  - Research Site 13, Sugar Land, Texas
  - Research Site 25, Victoria, Texas
  - Research Site 15, Bountiful, Utah
  - Research Site 35, St. George, Utah
  - Research Site 10, Manassas, Virginia
- Canada (6):
  - Research Site 20, Victoria, British Columbia
  - Research Site 7, London, Ontario
  - Research Site 6, Chicoutimi, Quebec
  - Research Site 5, Montreal, Quebec
  - Research Site 19, Québec, Quebec
  - Research Site 4, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No